CLINICAL TRIAL: NCT04121637
Title: To Investigate the Effect of Aerobic Exercise on Neurophysiological Values and Functionality in Individuals With Multiple Sclerosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Firat University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FiratUniversity
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; FNDC5; Irisin Hormone; Aerobic Exercise; EMG: Axonal Abnormality
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Control group Working group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the person who will make the analysis will not know the applications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise+Frenkel coordination Study group (Experimental): Patients will be given Frenkel Coordination exercises (4 different exercises 4-5 repetitions depending on the individual's functional and motor status) 3 times a week for 6 weeks. There will be a 1 minute break between each exercise set. Following this, an aerobic exercise of 30 minutes will be performed on the bicycle ergometer with electronic brake. Subjects will be advised not to do any exercise two days before or on that day and to eat only a light meal at least two hours before the test. The intensity of the exercise will be adjusted based on maximum oxygen consumption (VO2 max) specific to each individual.
  Interventions: Other: Aerobic Exercise; Other: Frenkel coordination exercises
- Frenkel coordination exercise group - Control group (Active Comparator): Patients will be given Frenkel Coordination exercises (4 different exercises 4-5 repetitions depending on the individual's functional and motor status) 3 times a week for 6 weeks. There will be a 1 minute break between each exercise set.
  Interventions: Other: Frenkel coordination exercises

INTERVENTIONS:
Other: Aerobic Exercise — Each exercise session;
  * 5 min warm-up = 30% of VO2 max
  * 20 min exercise = 50-60% of VO2 max
  * 5 minutes cooling in the form. The goal of aerobic exercise is to increase physical capacity, which is represented by maximum oxygen uptake (VO2max) and mechanical power generated during exercise. Training programs should be conducted at least 2 to 3 times per week (60-80% maximum work rate or 60% VO2max) for 30 to 60 minutes at moderate concentrations. These programs are effective in increasing aerobic capacity and power output in MS.
  Arms: Aerobic exercise+Frenkel coordination Study group
Other: Frenkel coordination exercises — Patients will be given Frenkel Coordination exercises (4 different exercises 4-5 repetitions depending on the individual's functional and motor status) 3 times a week for 6 weeks. 1 minute break between each exercise set

SUMMARY:
Multiple sclerosis (MS), a chronic inflammatory disease of the central nervous system, is characterized by myelin, oligodendrocytes and axon damage.

Physical exercises can be beneficial to patients, reduce fatigue and improve their strength, endurance and quality of life. Exercise has the potential to improve and / or preserve functionality, aerobic condition, strength, fatigue, health-related quality of life, depression, and cognition in MS patients. It has been reported that aerobic exercise increases muscle strength and endurance in peak oxygen intake and decreases fatigue and improves activity level, balance and walking patterns.

It is important to control the problems caused by ataxia in MS patients, to improve balance and postural reactions and to increase proximal muscle and trunk stabilization. For this purpose, movements are voluntarily and graded. Progress in exercises is achieved by making changes in the speed, width and complexity of movement. However, Frenkel Coordination exercises for extremity ataxia are usually included in the physiotherapy and rehabilitation program.

Little is known about the role and function of the iris in the nervous system with the discovery of Irisin and its precursor protein FNDC5. Evidence that the plasma level of iris increases during physical exercise suggests that it may also have beneficial and neuroprotective effects in the brain. Increased physical exercise has been shown to be associated with FNDC5 expression and ultimately more secretion of the iris.

The effect of elevated plasma iris levels after aerobic exercise on functionality in MS patients is unknown. Moon et al. Observed that cellular proliferation in mouse hippocampus cells was dose-dependent due to iris. In spraque dawley-type male rats, the presence of significant iris in the myelin sheath of the skeletal muscle shows that this tissue is an important source of iris. Based on these findings, it is thought that exercise-induced iris, which is an important cause of disability in MS, may have beneficial effects on the recovery of normal function in these patients. Whether iris affects nerve conduction velocity will be determined by electromyography analysis before and after aerobic exercise. In addition, the relationship between aerobic exercise and motor and sensory function and iris will be investigated and evaluated with functional tests.

DETAILED DESCRIPTION:
Purpose of the research:

The aim of this study is to investigate the effect of aerobic exercise on neurophysiological values and functionality in individuals with multiple sclerosis.

The aim of this study is to determine whether aerobic exercise has positive effects on neurophysiological values and functionality in MS patients and to investigate this in a multidisciplinary and multidisciplinary manner.

Materials and Methods:

Patients with MS who were referred to the physiotherapy and rehabilitation program by the Physical Medicine and Rehabilitation specialist at Fırat University Training and Research Hospital will be included in the study.

In this study, patients with MS will be divided into two groups by stratified randomization method. Stratification will be performed in the early period of MS (EDSS 0.5-2.5) and in the late period of MS (EDSS 3-5.5). For a total of 18 sessions, only Frenkel Coordination exercises will be done to the control group, and Frenkel Coordination exercises and aerobic exercise will be applied to the study group.

Physiotherapy and Rehabilitation Program Control Group: Patients will receive Frenkel Coordination exercises (4 different exercises 4-5 repetitions depending on the individual's functional and motor status) for 6 weeks. There will be a 1 minute break between each exercise set.

Study Group: Patients will receive Frenkel Coordination exercises (4 different exercises 4-5 repetitions depending on the individual's functional and motor status) for 6 weeks. There will be a 1 minute break between each exercise set. Following this, an aerobic exercise of 30 minutes will be performed on the bicycle ergometer with electronic brake. Subjects will be advised not to do any exercise two days before or on that day and to eat only a light meal at least two hours before the test. The intensity of the exercise will be adjusted based on maximum oxygen consumption (VO2 max) specific to each individual.

Each exercise session;

* 5 min warm-up = 30% of VO2 max
* 20 min exercise = 50-60% of VO2 max
* 5 minutes cooling in the form. The goal of aerobic exercise is to increase physical capacity, which is represented by maximum oxygen uptake (VO2max) and mechanical power generated during exercise. Training programs should be conducted at least 2 to 3 times per week (60-80% maximum work rate or 60% VO2max) for 30 to 60 minutes at moderate concentrations. These programs are effective in increasing aerobic capacity and power output in MS (16).

Oxygen consumption (VO2), exhaled carbon dioxide (VCO2), minute ventilation (VE), respiratory rate (RR), respiration change rate (RER) and oxygen saturation (SaO2) will be recorded.

Evaluation Protocol:

Electromyography (EMG), max VO2 values and iris levels are analyzed before and after treatment and scales and questionnaires will be applied to evaluate the functional levels.

Within the scope of EMG evaluation, motor and sensory conduction studies of ulnar and median nerve in upper extremity, peroneal and tibial nerve in lower extremity, F response and H-reflex study in motor nerves, sensory conduction study of sural nerve in lower extremity are planned. H reflex is a monosynaptic reflection carried by 1a sensory fibers that synapse with alpha motor neuron. Response F shows the repeated discharges of alpha motor neurons and is a test used for the evaluation of diseases that cause transmission slowdown.

The VO2 max measurement will be performed using the incremental exercise test to determine the maximum aerobic capacity. After resting for 5 minutes (sitting on the ergometer), patients will be asked to start cycling on the ergometer starting at 25W. The load will be increased by 25W every 3 minutes until depletion. Subjects will be encouraged to continue the exercise as much as possible orally. Oxygen consumption (VO2), exhaled carbon dioxide (VCO2), minute ventilation (VE), respiration rate (RR), respiration change rate (RER), oxygen saturation (SaO2) and heart rate will be recorded. In the statistical analysis, only VO2 max values will be examined.

For the analysis of the level of iris, blood samples will be taken from gel biochemistry tubes as appropriate for the analyzes to be performed from the patients at the end of the aerobic capacity assessment. Blood samples will be separated by centrifugation at 3000rpm for 10min and the obtained sera will be placed in small portions in ependorf tubes and stored at -80 ° C until analysis. Irisin levels will be studied using commercial ELISA (enzyme-linked immunosorbent assay) kits in accordance with the kit user manual.

Multiple Sclerosis Functional Composite (MSFC), Ataxia Assessment and Rating Scale (SARA), Modified Borg Scale (MBS) to determine the effect of aerobic exercise on functionality in individuals with MS , Fatigue Impact Scale (FIS), Leeds Multiple Sclerosis Quality of Life Scale (Leeds Multiple Sclerosis Quality of L)

ELIGIBILITY:
Inclusion Criteria:

* EDSS score in the range of 0.5-5.5,
* Patients with relapsing-remitting type MS
* Patients diagnosed with MS who did not receive steroid therapy or were discontinued 3 months before starting the study.

Exclusion Criteria:

* Has an acute MS attack or has a history of attacks in the last 3 months,
* Have orthopedic or systemic problems to prevent participation in the exercises,
* Another known neuromuscular disorder other than MS,
* Immunomodulatory therapy started in the last 6 months,
* Have visual involvement or diplopia,
* Upper spasticity of lower limbs (Ashworth score 3 or 4),
* Patients with cardio-pulmonary problems that would prevent their participation in the exercise.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-10-21 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Physiological - Irisin Hormone | 8 mounth
  For the analysis of the level of iris, blood samples will be taken from gel biochemistry tubes as appropriate for the analyzes to be performed from the patients at the end of the aerobic capacity assessment. Blood samples will be separated by centrifugation at 3000rpm for 10min and the obtained sera will be placed in small portions in ependorf tubes and stored at -80 ° C until analysis. Irisin levels will be studied in accordance with the kit user manual using commercial ELISA (enzyme-linked immunosorbent assay) kits
Neurophysiological - EMG | 8 mounth
  In the scope of EMG evaluation, the motor and sensory conduction studies of the ulnar and median nerve in the upper extremity, the peroneal and tibial nerves in the lower extremity, the F response and H-reflex study in the motor nerves, and the sensory conduction study of the sural nerve in the lower extremity are planned.
VO2 Max | 8 mounth
  The VO2 max measurement will be performed using the incremental exercise test to determine the maximum aerobic capacity. After resting for 5 minutes (sitting on the ergometer), patients will be asked to start cycling on the ergometer starting at 25W. The load will be increased by 25W every 3 minutes until depletion.

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composites (MSFC) | 8 mounth
  Multiple Sclerosis Functional Composites (MSFC) was developed by the National MS Society's Clinical Outcomes Assessment Task Force. Objective assessment of functional disability score and help to maintain the standard of patient follow-up. It consists of 25 Step Walk Test, 9 Hole Peg Test, Step Auditory Serial Addition Test (PASAT) subtests. PASAT is used to measure the speed of auditory information processing, computational skills and attention from executive functions. It has two forms, A and B, and is performed with a standard voice recording. Each form has two subtests. In the first subtest, the numbers are repeated at three-second intervals, and the patient is expected to add the next number he heard. Each time, the patient must add the previous and the new number. 9 Perforated Peg Test is a test that measures upper extremity functions (hand and arm) and motor speed.
Ataxia Scale (SARA) | 8 mounth
  The Ataxia Scale (SARA) is a scale used to assess ataxia including clinical dysfunction, limb movements, kinetic functions, posture and gait disorders, speech and oculomotor disorders. SARA subscores are posture and gait, speech, kinetic functions of the extremities
Leeds Multiple Sclerosis Quality of Life Scale (LMSQoL) | 8 mounth
  The Leeds Multiple Sclerosis Quality of Life Scale (LMSQoL) was developed to assess the quality of life of individuals with MS. The eight-item form of this scale is directed towards fatigue, loneliness, energy, health concerns, family relationships, appearances, other people's attitudes, and the future. It is stated that LMSQoL is sensitive and reliable for the studied population and it is fast and easy to use in the clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer ÇETİŞLİ KORKMAZ, Principal Investigator — Pamukkale University; Zübeyde ERCAN, Principal Investigator — Firat University; Gökhan ALKAN, Principal Investigator — Firat University; Murat GÖNEN, Principal Investigator — Firat University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frohman EM, Racke MK, Raine CS. Multiple sclerosis--the plaque and its pathogenesis. N Engl J Med. 2006 Mar 2;354(9):942-55. doi: 10.1056/NEJMra052130. No abstract available. PMID 16510748
- [Background] Lassmann H, Bruck W, Lucchinetti CF. The immunopathology of multiple sclerosis: an overview. Brain Pathol. 2007 Apr;17(2):210-8. doi: 10.1111/j.1750-3639.2007.00064.x. PMID 17388952
- [Background] Dalgas U, Stenager E. Progressive resistance therapy is not the best way to rehabilitate deficits due to multiple sclerosis: no. Mult Scler. 2014 Feb;20(2):141-2. doi: 10.1177/1352458513513060. No abstract available. PMID 24493702
- [Background] Rietberg MB, Brooks D, Uitdehaag BM, Kwakkel G. Exercise therapy for multiple sclerosis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003980. doi: 10.1002/14651858.CD003980.pub2. PMID 15674920
- [Background] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230
- [Background] Petajan JH, Gappmaier E, White AT, Spencer MK, Mino L, Hicks RW. Impact of aerobic training on fitness and quality of life in multiple sclerosis. Ann Neurol. 1996 Apr;39(4):432-41. doi: 10.1002/ana.410390405. PMID 8619521
- [Background] Sarova-Pinhas I, Achiron A, Gilad R, Lampl Y. Peripheral neuropathy in multiple sclerosis: a clinical and electrophysiologic study. Acta Neurol Scand. 1995 Apr;91(4):234-8. doi: 10.1111/j.1600-0404.1995.tb06996.x. PMID 7625146
- [Background] Ayromlou H, Mohammad-Khanli H, Yazdchi-Marandi M, Rikhtegar R, Zarrintan S, Golzari SE, Ghabili K. Electrodiagnostic evaluation of peripheral nervous system changes in patients with multiple sclerosis. Malays J Med Sci. 2013 Jul;20(4):32-8. PMID 24043994
- [Background] Armutlu K, Karabudak R, Nurlu G. Physiotherapy approaches in the treatment of ataxic multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2001;15(3):203-11. doi: 10.1177/154596830101500308. PMID 11944742
- [Background] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023
- [Background] Wrann CD, White JP, Salogiannnis J, Laznik-Bogoslavski D, Wu J, Ma D, Lin JD, Greenberg ME, Spiegelman BM. Exercise induces hippocampal BDNF through a PGC-1alpha/FNDC5 pathway. Cell Metab. 2013 Nov 5;18(5):649-59. doi: 10.1016/j.cmet.2013.09.008. Epub 2013 Oct 10. PMID 24120943
- [Background] Moon HS, Dincer F, Mantzoros CS. Pharmacological concentrations of irisin increase cell proliferation without influencing markers of neurite outgrowth and synaptogenesis in mouse H19-7 hippocampal cell lines. Metabolism. 2013 Aug;62(8):1131-6. doi: 10.1016/j.metabol.2013.04.007. Epub 2013 May 7. PMID 23664146
- [Background] Novelle MG, Contreras C, Romero-Pico A, Lopez M, Dieguez C. Irisin, two years later. Int J Endocrinol. 2013;2013:746281. doi: 10.1155/2013/746281. Epub 2013 Nov 5. PMID 24298283
- [Background] Aydin S, Kuloglu T, Aydin S, Eren MN, Celik A, Yilmaz M, Kalayci M, Sahin I, Gungor O, Gurel A, Ogeturk M, Dabak O. Cardiac, skeletal muscle and serum irisin responses to with or without water exercise in young and old male rats: cardiac muscle produces more irisin than skeletal muscle. Peptides. 2014 Feb;52:68-73. doi: 10.1016/j.peptides.2013.11.024. Epub 2013 Dec 15. PMID 24345335
- [Background] Briken S, Rosenkranz SC, Keminer O, Patra S, Ketels G, Heesen C, Hellweg R, Pless O, Schulz KH, Gold SM. Effects of exercise on Irisin, BDNF and IL-6 serum levels in patients with progressive multiple sclerosis. J Neuroimmunol. 2016 Oct 15;299:53-58. doi: 10.1016/j.jneuroim.2016.08.007. Epub 2016 Aug 5. PMID 27725121
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Harvey L, Smith AD, Jones RJP. The effect of weighted leg raises on quadriceps strength, EMG parameters and functional activities in people with multiple sclerosis. 1999;85(3):154-61.
- [Background] Schulz KH, Gold SM, Witte J, Bartsch K, Lang UE, Hellweg R, Reer R, Braumann KM, Heesen C. Impact of aerobic training on immune-endocrine parameters, neurotrophic factors, quality of life and coordinative function in multiple sclerosis. J Neurol Sci. 2004 Oct 15;225(1-2):11-8. doi: 10.1016/j.jns.2004.06.009. PMID 15465080
- [Background] Tsuchiya Y, Mizuno S, Goto K. Irisin response to downhill running exercise in humans. J Exerc Nutrition Biochem. 2018 Jun 30;22(2):12-17. doi: 10.20463/jenb.2018.0011. PMID 30149421
- [Background] Fischer JS, Rudick RA, Cutter GR, Reingold SC. The Multiple Sclerosis Functional Composite Measure (MSFC): an integrated approach to MS clinical outcome assessment. National MS Society Clinical Outcomes Assessment Task Force. Mult Scler. 1999 Aug;5(4):244-50. doi: 10.1177/135245859900500409. PMID 10467383
- [Background] Fischer JS, Jak A, Kniker J, Rudick R, Cutter GJNYNMSS. Multiple Sclerosis Functional Composite (MSFC): administration and scoring manual. 2001.
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946
- [Background] Armutlu K, Keser I, Korkmaz N, Akbiyik DI, Sumbuloglu V, Guney Z, Karabudak R. Psychometric study of Turkish version of Fatigue Impact Scale in multiple sclerosis patients. J Neurol Sci. 2007 Apr 15;255(1-2):64-8. doi: 10.1016/j.jns.2007.01.073. Epub 2007 Mar 6. PMID 17337007
- [Background] Polat C, Tulek Z, Kurtuncu M, Eraksoy M. Validity and Reliability of the Turkish Version of the Monitoring My Multiple Sclerosis Scale. Noro Psikiyatr Ars. 2017 Jun;54(2):131-136. doi: 10.5152/npa.2016.12694. Epub 2017 Jan 19. PMID 28680310
- [Background] Hisli N. Beck Depresyon Olcegi'nin bir Turk ornekleminde gecerlilik ve guvenilirligi. Psikoloji Dergisi 1988; 6:118-122.